CLINICAL TRIAL: NCT06554002
Title: The Acute-postprandial and Long-term Effects of Different Types of Carbohydrate on Human Health and Blood Glucose Management
Brief Title: Acute and Long-term Health Effects of Various Carbohydrates on Blood Glucose Management in Humans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Singapore Institute of Food and Biotechnology Innovation (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2017/00558
Record Dates: First submitted 2024-07-26; First posted 2024-08-14 (Actual); Last update posted 2024-08-14 (Actual); Status verified 2024-08

CONDITIONS: Nutrition, Healthy
Keywords: resistant dextrin; glycaemic control; insulin sensitivity
MeSH Terms: conditions — Insulin Resistance | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: Crossover assignment. Single-blinded, randomized, controlled, parallel arm trial with each participant block-randomized into either control or treatment group
Masking Description: Single-blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Experimental): Flavoured beverage powder with 3g glucose, twice a day
  Interventions: Other: Control
- Treatment (Experimental): Flavoured beverage powder with 20g resistant dextrin, twice a day
  Interventions: Other: Treatment

INTERVENTIONS:
Other: Control — Participants will be asked to consume glucose on a daily basis (twice per day) for the entire 8 weeks. The supplement will be packed in sachets, and it can be dissolved in water to be consumed as a beverage. Two sachets will be consumed daily.
  Arms: Control
Other: Treatment — Participants will be asked to consume a resistant dextrin on a daily basis (twice per day) for the entire 8 weeks. The test supplement will be packed in sachets, and it can be dissolved in water to be consumed as a beverage. Two sachets will be consumed daily.
  Arms: Treatment

SUMMARY:
Dietary fibre, especially soluble fibre, has several health benefits such as lowering the risks for cardiovascular disease, stroke, diabetes, obesity, and gastrointestinal diseases. Resistant dextrin is a non-viscous soluble fibre, can be introduced quite easily in foods or as drinks, and it is well tolerated. This study aims to investigate if daily supplementation of habitual diets with resistant dextrin over 8 weeks affect glycaemic control via insulin sensitivity, intestinal fermentation, energy expenditure and fat oxidation in adults with increased risk for type 2 diabetes. The primary outcome is the effect on glycaemic control (fasting glucose, insulin, insulin sensitivity and 24 hour glycaemic response from CGMS). The secondary outcomes are the effects on fasting lipids, energy expenditure and fuel utilization in a whole room calorimeter and appetite regulation.

DETAILED DESCRIPTION:
Dietary fibre has several health benefits such as lowering the risks for cardiovascular disease, stroke, diabetes, obesity, and gastrointestinal diseases. Dietary fibre intake has regularly been reported to be below the daily recommended levels. Based on the 2010 National Nutrition Survey, 21% of Singaporeans did not meet the recommended daily intake of dietary fibre. While increasing fruit and vegetables intake remains the primary strategy to promote fibre intake, an alternative is to supplement a daily diet with dietary fibre, especially soluble fibre, to improve health.

Resistant dextrin is a non-viscous soluble fibre that exhibits prebiotic properties and it has been shown to alter gastrointestinal ecology. Emerging evidence suggests that resistant dextrin reduced insulin resistance in both healthy individuals and adults with type 2 diabetes, resulting in better blood glucose control. In term of its cardio-protective effects, resistant dextrin has also been shown to lower blood cholesterol levels and reduced inflammation biomarkers. Resistant dextrin has also been shown to suppress hunger and increase satiety, leading to reduced daily energy intake and greater body weight loss.

To date, evidence from clinical trials, notably among Asians is still insufficient to make dietary recommendations. In addition, the possibility of short-chain fatty acid production in stimulating diet-induced thermogenesis and fat oxidation has not been explored. These are the novel aspects that our proposed study aims to investigate.

ELIGIBILITY:
Inclusion Criteria:

* 21 to 60 years old
* Group A: 21 - 25 kg/m2, with first degree family history of type 2 diabetes, or Group B: 23 - 30 kg/m2, with waist circumference >85 cm for males and >82 cm for females

Exclusion Criteria:

* • Consume fibre supplements or any other supplements that is likely to interfere with study outcomes

  * Have any major organ dysfunction (e.g. cardiovascular, respiratory, hepatic, renal, gastrointestinal) that may influence taste, olfaction, appetite, digestion, metabolism, absorption or elimination of test foods, nutraceutical or drug
  * Smoking
  * Have any metabolic diseases (e.g. diabetes, hypertension)
  * Have medical conditions and/or taking medications known to affect glycaemia (e.g. glucocorticoids, thyroid hormones, thiazide diuretics)
  * Have glucose-6-phosphate dehydrogenase (G6PD) deficiency
  * Have any severe food allergy (e.g. anaphylaxis to peanuts), or any other known food allergy/intolerance
  * Have active Tuberculosis (TB) or currently receiving treatment for TB
  * Have any known Chronic infection or known to suffer from or have previously suffered from or is a carrier of Hepatitis B Virus (HBV), Hepatitis C Virus (HCV), Human Immunodeficiency Virus (HIV)
  * A team member of the study or their immediate family members (i.e. spouse, parent, child, or sibling, whether biological or legally adopted)
  * Enrolled in a concurrent research study judged not to be scientifically or medically compatible with the study of the CNRC.
  * Intentionally restricting food intake
  * Have poor veins impeding venous access
  * Have any history of severe vasovagal syncope (blackouts or near faints) following blood draws
  * Have claustrophobia

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 98 (Actual)
Dates: Start 2019-08-14 (Actual); Primary Completion 2023-08-14 (Actual); Study Completion 2023-08-14 (Actual)

PRIMARY OUTCOMES:
Glucose will be measured from fasting blood samples that will be collected at baseline (0 week), follow up visit (at 4 weeks) and at the end of the intervention (at 8 weeks). | Mid intervention visit on Week 4
  Fasting blood biochemistry from 14mL of venous blood sample collected via venipuncture.
Insulin will be measured from fasting blood samples that will be collected at baseline (0 week), follow up visit (at 4 weeks) and at the end of the intervention (at 8 weeks). | Mid intervention visit on Week 4
  Fasting blood biochemistry from 14mL of venous blood sample collected via venipuncture.
Insulin sensitivity will be measured from fasting blood samples that will be collected at baseline and final visit. | Mid intervention visit on Week 4
  Fasting blood biochemistry from 14mL of venous blood sample collected via venipuncture.
24 hour glycaemic response will measured in all participants during the baseline and at the end of the intervention (at 8 weeks). | Inserted on the Baseline visit (0 week) (Days 1-3) and Final visit (8 week) (Days 1-3)
  On Day 1 of the baseline and final test visits, participants will come to the laboratory in the evening (1600h) for continuous glucose monitoring system, CGMS (IPro®2, Medtronic, USA) insertion.

SECONDARY OUTCOMES:
Lipids will be measured measured from fasting blood samples that will be collected at baseline (0 week), follow up visit (at 4 weeks) and at the end of the intervention (at 8 weeks). | Mid intervention visit on Week 4
  Fasting blood biochemistry from 14mL of venous blood sample collected via venipuncture.
In a subset of 10 participants per study arm, energy expenditure will be measured in a whole room calorimeter on the baseline visit (0 week) and final visit (8 week), | On Day 2 of baseline visit (0 week) for 9 hours
  Energy expenditure measured in a whole room calorimeter (WRC).
Subjective appetite sensations collected before breakfast and lunch, and 4 hours postprandially at every half an hour, using validated 100mm visual analog scale questionnaires. | Before breakfast and lunch, and 4 hours postprandial breakfast and lunch, obtained every half an hour. VAS conducted on Day 2 of baseline (0 week) and final visit (8 week).
  Subjective appetite sensations collected using validated 100mm visual analog scale questionnaires. Four questions on hunger, fullness, desire to eat, prospective consumption. Questions anchored at 0 mm being the "least" and at 100 mm being "most". For example, for prospective consumption " How much food do you think you can eat now?", at 0mm (nothing at all) to 100 mm (a large amount). Results captured electronically using the software AVAS (available at: http://www.nrlc-group.net/software/AdaptiveVisual.php).

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Nutrition Research Centre (CNRC), Singapore, Singapore